CLINICAL TRIAL: NCT02877355
Title: Investigation of the Effect of Upper Gastrointestinal Disease on the Pharmacokinetics of Oral Semaglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4267; 2015-004534-10 (EudraCT Number); U1111-1175-5246 (Other: WHO)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — All subjects will receive 3 mg oral semaglutide for five days followed by 7 mg oral semaglutide for five days

SUMMARY:
This trial is conducted in Europe. The aim of this trial is, to investigate the effect of upper gastrointestinal disease on the pharmacokinetics (the exposure of the trial drug in the body) of oral semaglutide in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-80 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 18.5-39.9 kg/m^2 (both inclusive)
* Subjects diagnosed clinically with type 2 diabetes mellitus for at least 180 days prior to the first screening visit
* For subjects with upper gastrointestinal (GI) disease: Diagnosed with chronic gastritis and/or gastroesophageal reflux disease (GERD) at screening

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method (adequate contraceptive measures as required by local regulation or practice). (Highly effective contraceptive methods are considered those with a failure rate less than 1% undesired pregnancies per year including surgical sterilisation, hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence or a surgically sterilised partner)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Unable or unwilling to refrain from smoking during the in-patient periods
* Any blood draw in excess of 50 mL in the past 30 days, or donation of blood or plasma in excess of 400 mL within 90 days of the first screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration-time curve | From 0 to 24 hours after the 10th dosing

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | From 0 to 24 hours after the 10th dosing
Area under the SNAC plasma concentration-time curve | During a dosing interval (0 to 24 hours) at steady state
Maximum observed SNAC plasma concentration | During a dosing interval (0 to 24 hours) at steady state

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Overgaard RV, Navarria A, Ingwersen SH, Baekdal TA, Kildemoes RJ. Clinical Pharmacokinetics of Oral Semaglutide: Analyses of Data from Clinical Pharmacology Trials. Clin Pharmacokinet. 2021 Oct;60(10):1335-1348. doi: 10.1007/s40262-021-01025-x. Epub 2021 May 10. PMID 33969456
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com